CLINICAL TRIAL: NCT04599270
Title: Efficiency of Prevention Program Dedicated to Addictive Behaviors (PREVENTURE) of Vulnerable Teenagers
Acronym: PREVADO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC20.0114
Record Dates: First submitted 2020-10-12; First posted 2020-10-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Addiction, Alcohol; Addiction, Substance
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Teenager encounter psychologist for conduct a Substance Use risk Personality Scale (SURPS) assessment to identify personality characteristics that represent a risk for the development of problematic substance use. Only adolescents with at-risk personality traits according to the SURPS will be randomized for further assessment.
  If adolescent have not risk personality traits, the patient will go out of the study.
  If adolescent have risk personality traits, other tests and scales will be performed to study the intensivity of dependance of substance use and the patient will be randomized.
  If he is randomized in intervention group, the patient will follow PREVENTURE program (2 session of 90 min by videoconference), within 3 months after inclusion and will be contacted by phone by the psychologist at 1, 3, 6 and 12 month after sessions to answer the same tests and scales.
  Interventions: Other: PREVENTURE Program
- Control group (Active Comparator): Teenager encounter psychologist for conduct a Substance Use risk Personality Scale (SURPS) assessment to identify personality characteristics that represent a risk for the development of problematic substance use. Only adolescents with at-risk personality traits according to the SURPS will be randomized for further assessment.
  If adolescent have not risk personality traits, the patient will go out of the study.
  If adolescent have risk personality traits, other tests and scales will be performed to study the severity of substance use disorders and the patient will be randomized.
  If he is randomized in control group, the patient will follow routine care and will be contacted by phone by the psychologist at 1, 3, 6 and 12 month after inclusion to answer the same tests and scales.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: PREVENTURE Program — Adolescents will be follow PREVENTURE program (2 session of 90 min).
  Arms: Intervention group
Other: Routine care — Adolescents will be follow routine care
  Arms: Control group

SUMMARY:
At the age of 17, in Brittany, 94.9% of adolescents have experimented alcohol consumption 78.1% within a month and 25.5% report repeated episodes of Intensive Punctual Alcohol. Among the potential explanatory factors of this worrying epidemiology, social and cultural factors induce a social valuation of alcohol consumption and drunkenness. There are also individual vulnerability factors, particularly important in adolescence between experimentation and the transition to regular use or even to alcohol use disorders. Despite the extent of the damage, there is currently little reliable data on effective primary prevention strategies for dealing with addictive behavior. Many prevention programs target age range in school settings, to delay or reduce use of psychoactive substances.

A meta-analysis on the impact of this prevention programs in school settings, concluded that most interventions are associated with no or little impact with respect to the goal of reducing psychoactive substances with teenagers.

Among existing programs, "PREVENTURE" has been evaluated in 5 trials with high-risk teenagers identified in schools settings, in different countries (Canada, Europe). The results show a clear and robust effect on reducing alcohol consumption. This program has not been tested outside the school setting and a recent review mention the need to make this program more accessible by targeting vulnerable groups and studying the impact of this program on this population.

The PREVADO study is a prospective, controlled, randomised, open-label study. After inclusion, the adolescent completes the questionnaire SURPS (Substance Use Risk Profile Scale).

The SURPS is self-report questionnaire that assesses four well-validated personality risk factors for substance misuse (Impulsivity, Sensation Seeking, Anxiety Sensitivity, and Hopelessness). There is a 23-item to which adolescents are asked to respond using a 4-point Likert scale ranging from "strongly agree" to "strongly disagree" : Hopelessness (7 items), Anxiety Sensitivity (5 items), Impulsivity (5 items), and Sensation Seeking (6 items).

Adolescents will be randomized into 2 groups (stratification on the 4 predominant risk personality types from the SURPS (Substance Use Risk Profile Scale) and on the recruitment modality) :

* Intervention group : teenagers follow the "PREVENTURE" program and routine cares
* Control group : teenagers follow routine cares

ELIGIBILITY:
Inclusion Criteria:

* Aged between 14 and 17 years old
* Patient consulting in one of the participating centres or referred by a school doctor
* Patient who has had at least one previous experience with alcohol (at least 1 standard unit of alcohol, once in their lifetime)
* Having access to an internet network and a computer, tablet or telephone
* Written and informed consent of the parents and the teenager

Exclusion Criteria:

* Refusal to participate in the study
* Moderate to Severe Adolescent Substance Use Disorders (other than smoking)
* Decompensated current psychiatric disorders in adolescents
* Already followed for severe use disorders and/or severe psychiatric disorders
* Nonunderstanding of the french language

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Intensive Punctual Alcohol | Month 6
  The primary endpoint will be the occurrence of at least one Intensive Punctual Alcohol (at least 5 unit standard of alcohol at one time) within the last month (assessed at 6 months) as measured by the Alcohol Timeline Followback (ATLFB). The TLFB is a method for assessing recent drinking behavior. It involves asking clients to retrospectively estimate their daily alcohol consumption over a time period for 30 days prior to the interview.

SECONDARY OUTCOMES:
Evaluation of substance use | Day 0, Month 1, Month 3, Month 6 and Month 12
  Criteria for assessing alcohol, tobacco or cannabis use: experimentation / use within the month / regular (more than 10 times a month) as measured by the Alcohol Timeline Followback (ATLFB). The TLFB is a method for assessing recent drinking behavior. It involves asking clients to retrospectively estimate their daily alcohol consumption over a time period for 30 days prior to the interview.
Evaluation of alcohol consumption type | Day 0, Month 6 and Month 12
  Alcohol consumption type will be evaluated by Alcohol Use Disorders Identification Test (AUDIT) scale. AUDIT is a 10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. A score of 8 or more is considered to indicate hazardous or harmful alcohol use.
Evaluation of tobacco consumption type | Day 0, Month 6 and Month 12
  Tobacco consumption type will be evaluated by Hooked on Nicotine Checklist (HONC) scale. HONC is a 10-item instrument used to determine the onset and strength of tobacco dependence. A positive response to any HONC item signals a loss of autonomy and the onset of dependence.
Evaluation of cannabis consumption type | Day 0, Month 6 and Month 12
  Cannabis consumption type will be evaluated by Cannabis Abuse Screening Test (CAST) scale. CAST is a 6-item screening tool to assess cannabis consumption and cannabis-related problems. A score between 3 and 6 means a low risk and greater than or equal to 7 means a high risk of addiction.
Evaluation of alcohol and drugs consumption type | Day 0, Month 6 and Month 12
  Alcohol and drugs consumption type will be evaluated by ADOlescents et Substances Psyhco-Actives (ADOSPA) scale. ADOSPA scale is a simple test for the early detection of risky and harmful use of alcohol or drugs among young people. It consists of 6 items. A score higher than 3 indicates high risk.
Evaluation of anxiety and depression | Day 0, Month 1, Month 3, Month 6 and Month 12
  Anxiety and depression will be evaluated by Adolescent Depression Rating Scale (ADRS). Adolescent depression rating scale (ADRS) assesses depression in adolescents in 10 items. The items measure insomnia, anxiety, sadness and fatigability. If ADRS score is less than 4 : low risk of depression, between 4 and 8 : moderate risk of depression and superior than 8 : significant risk of depression.
Evaluation of alcohol-related harm | Day 0, Month 1, Month 3, Month 6 and Month 12
  Collected negative events related to alcohol consumption in the past month assessed at at medical interview.
Evaluation of quality of life | Day 0, Month 1, Month 3, Month 6 and Month 12
  The quality of life will be evaluated by Pediatric Quality of Life InventoryTM (PedsQL) scale. 3 scores will be calculated : psychosocial health summary score (average score of 15 items), physical health summary score (average score of 8 items) and the total score (average score of all items). Scores are between 0 and 100% and the higher scores indicate better Health-Related Quality of Life.
Evaluation of acceptability of the study | Day 0, Month 1, Month 3, Month 6 and Month 12
  The evaluation of acceptability of the study by the adolescents was evaluated by the participation rate the adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Morgane GUILLOU - LANDREAT, Dr, Principal Investigator — CHRU Brest
Locations (5):
- France (5):
  - Loik JOUSNI, Brest
  - Morgane GUILLOU - LANDREAT, Brest
  - Pascale ROZEC, Landerneau
  - Catherine SIMON, Morlaix
  - Benoit SCHRECK, Nantes

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 51 month and ending 15 years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Guillou-Landreat M, Tahmazov E, Benoit S, Grall-Bronnec M, Conrod P, Livet A, Nowak E, Le Reste J-. The efficacy of a targeted PREVENTION programme for addictive behaviour (PREVENTURE) among vulnerable ADOlescents in France - study procotol. BMC Public Health. 2021 Apr 23;21(1):783. doi: 10.1186/s12889-021-10795-9. PMID 33892682